CLINICAL TRIAL: NCT01694433
Title: Innate Immunity in Acne Vulgaris
Brief Title: "Clinical Trial to Determine the Efficacy of Vitamin D for Acne Therapy"
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Jenny Kim, MD, PhD, Professor of Medicine/Dermatology, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01AR053542-01A2 (NIH); 1R01AR053542-01A2 (NIH)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Calcipotriene Cream (Experimental): The Calcipotriene Cream will be supplied as 1g daily use individual tubes to be used 2x/day (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Calcipotriene
- Placebo (Placebo Comparator): The Placebo Cream will be supplied as 1g daily use individual tubes to be used 2x/day (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcipotriene — 1g daily BID
  Other Names: Dovonex; Vitamin D cream
  Arms: Calcipotriene Cream
Drug: Placebo — 1g daily BID
  Other Names: Placebo cream manufactured to mimic calcipotriene
  Arms: Placebo

SUMMARY:
The purpose of this study is to study the effects of topical Vitamin D cream (Calcipotriene, also known as Dovonex) on acne. The information gained from this study may lead to new treatments for acne. In this study, Calcipotriene will be compared with a placebo, a cream that looks like Calcipotriene, but contains no active ingredients.

DETAILED DESCRIPTION:
This study will be a randomized, double-blinded, parallel group comparison of calcipotriene vs. placebo cream. Patients with acne will use calcipotriene or placebo cream 2x/day for 12 weeks and will be assessed at weeks 0, 2, 4, 8 and 12. Each group will have 24 subjects as calculated by power analysis. Three additional subjects for each group will be recruited for possible dropouts and total of 27 subjects will be recruited for each group. Primary endpoint (lesion count) and secondary endpoint (IGA- Investigator's Global Assessment) will be determined. Lesion counts will be assessed by one of the investigator physicians or nurse practitioner. Adverse effects including irritation, dry skin, inflammation and worsening of the lesions will be noted at each visit. Photographs will be taken to aid in assessing the clinical changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, of either gender and any racial/ethnic group
2. Subjects must have clinically evident mild to moderate acne vulgaris of the facial area, IGA scale, grade 2-4
3. Subjects must understand and sign the informed consent prior to participation
4. Subjects must be in generally good health
5. Subjects must be able and willing to comply with the requirements of the protocol

Exclusion Criteria:

1. Oral retinoid use within twelve months of entry into the study
2. Systemic acne therapies (oral antibiotics) within 30 days of entry into the study
3. Topical acne therapies (retinoids, antibiotics) within 14 days of entry into the study
4. Non-compliant patients
5. Pregnant or nursing women
6. Subjects with a significant medical history or concurrent condition that the investigator(s) feel is not safe for study participation
7. Subjects with hypercalcemia (hyperparathyroidism, kidney disease)
8. Subjects who cannot avoid excessive exposure to either natural or artificial sunlight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Kim, MD,PhD, Principal Investigator — UCLA Department of Medicine/Division of Dermatology and Nutrition
Locations (1):
- UCLA Dermatology, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcipotriene Cream: The Calcipotriene Cream supplied as 1g daily use individual tubes used 2x/day (once in the morning and once in the evening) for 12 weeks.
  Calcipotriene: 1g daily BID
- Placebo: The Placebo Cream supplied as 1g daily use individual tubes used 2x/day (once in the morning and once in the evening) for 12 weeks.
  Placebo: 1g daily BID
Period: Overall Study
Arm/Group | Calcipotriene Cream | Placebo
Started | 33 | 33
Baseline Visit | 33 | 32
Completed | 22 | 29
Not Completed | 11 | 4
Not completed — Adverse Event | 7 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Population: One enrolled participant withdrew from the Placebo arm prior to Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcipotriene Cream | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65
Inflammatory Lesion Count [Mean (Full Range); unit: Lesions] | 16.8 [0 to 59] | 11.7 [1 to 34] | 14.3 [1 to 59]
Non-inflammatory Lesion Count [Mean (Full Range); unit: Lesions] | 48.4 [4 to 440] | 38.4 [2 to 141] | 43.5 [4 to 440]
Total Lesion Count [Mean (Full Range); unit: Lesions] | 67.3 [13 to 452] | 50.1 [5 to 146] | 57.8 [5 to 452]
IGA at Baseline [Mean (Full Range); unit: score on a scale] — Investigator's Global Assessment (IGA) is a 5-point scale of acne severity, ranging from 0 (Clear) to 4 (Severe)
  score on a scale | 3.15 [2 to 4] | 3.06 [1 to 4] | 3.11 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Lesion Counts (Total, Inflammatory and Non-inflammatory)
Description: Lesion counts will be assessed by one of the investigator physicians or nurse practitioner.
Time Frame: Weeks 2, 4, 8 & 12
Population: The number of participants analyzed differ from overall number analyzed due to participant withdrawal or missed study visit.
Measure: Mean (Full Range); unit: Lesions
Arm/Group | Calcipotriene Cream | Placebo
Number analyzed (Participants) | 33 | 32
Lesions
  Inflammatory lesions at Week 2: number analyzed (Participants) | 30 | 31
  Inflammatory lesions at Week 2 | 18.4 [1 to 89] | 13.4 [0 to 66]
  Inflammatory lesions at Week 4: number analyzed (Participants) | 24 | 27
  Inflammatory lesions at Week 4 | 15.8 [0 to 66] | 9.9 [1 to 34]
  Inflammatory lesions at Week 8: number analyzed (Participants) | 24 | 29
  Inflammatory lesions at Week 8 | 12.1 [0 to 94] | 10.2 [0 to 31]
  Inflammatory lesions at Week 12: number analyzed (Participants) | 22 | 29
  Inflammatory lesions at Week 12 | 10.5 [0 to 37] | 7.0 [0 to 43]
  Non-inflammatory lesions at Week 2: number analyzed (Participants) | 30 | 31
  Non-inflammatory lesions at Week 2 | 30.9 [1 to 152] | 33.1 [0 to 131]
  Non-inflammatory lesions at Week 4: number analyzed (Participants) | 24 | 27
  Non-inflammatory lesions at Week 4 | 35.5 [3 to 299] | 34.4 [0 to 198]
  Non-inflammatory lesions at Week 8: number analyzed (Participants) | 24 | 29
  Non-inflammatory lesions at Week 8 | 22.1 [0 to 136] | 24.3 [0 to 110]
  Non-inflammatory lesions at Week 12: number analyzed (Participants) | 22 | 29
  Non-inflammatory lesions at Week 12 | 19.6 [0 to 78] | 20.2 [1 to 60]
  Total lesions at Week 2: number analyzed (Participants) | 30 | 31
  Total lesions at Week 2 | 51.0 [6 to 241] | 46.5 [2 to 158]
  Total lesions at Week 4: number analyzed (Participants) | 24 | 27
  Total lesions at Week 4 | 51.4 [0 to 299] | 44.3 [2 to 232]
  Total lesions at Week 8: number analyzed (Participants) | 24 | 29
  Total lesions at Week 8 | 34.2 [0 to 136] | 34.55 [1 to 134]
  Total lesions at Week 12: number analyzed (Participants) | 22 | 29
  Total lesions at Week 12 | 30.1 [0 to 78] | 27.24 [2 to 73]

2. Secondary Outcome: Acne Severity as Assessed With the Investigator's Global Assessment (IGA)
Description: Investigator's Global Assessment (IGA) is a 5-point scale of acne severity, ranging from 0 (Clear) to 4 (Severe)
Time Frame: Weeks 2, 4, 8 & 12
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Calcipotriene Cream | Placebo
Number analyzed (Participants) | 33 | 32
score on a scale
  IGA at Week 2: number analyzed (Participants) | 30 | 31
  IGA at Week 2 | 2.77 [1 to 4] | 2.9 [1 to 4]
  IGA at Week 4: number analyzed (Participants) | 24 | 27
  IGA at Week 4 | 2.83 [1 to 4] | 2.59 [1 to 4]
  IGA at Week 8: number analyzed (Participants) | 24 | 29
  IGA at Week 8 | 2.21 [1 to 4] | 2.48 [1 to 4]
  IGA at Week 12: number analyzed (Participants) | 22 | 29
  IGA at Week 12 | 2.23 [1 to 4] | 2.31 [1 to 4]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Calcipotriene Cream | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 18/33 | 19/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcipotriene Cream (N=33) | Placebo (N=32)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bug bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bump on eyelid (Eye disorders) | 0 (0) | 1 (1)
Common cold/allergy (Infections and infestations) | 10 (11) | 7 (8)
Facial dryness (Skin and subcutaneous tissue disorders) | 18 (22) | 5 (5)
Flu-like symptoms (General disorders) | 1 (1) | 2 (2)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1) | 1 (3)
GI Flu (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (3)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Facial irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Redness (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Sore Throat (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No